CLINICAL TRIAL: NCT04093076
Title: Dose-Ranging Study to Evaluate the Safety, Tolerability and Immunogenicity of INO-4500 in Combination With Electroporation in Healthy Volunteers in Ghana
Brief Title: Dose-ranging Study: Safety, Tolerability and Immunogenicity of INO-4500 in Healthy Volunteers in Ghana
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LSV-002
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Lassa Fever
Keywords: Healthy volunteer
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sponsor will be blinded up to Week 6; at that time the Sponsor will become group-level unblinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- INO-4500 Group A (Experimental): Participants will receive 1 ID injection of 1 mg/dose INO-4500 followed by EP using the CELLECTRA™ 2000 device.
  Interventions: Drug: INO-4500; Device: CELLECTRA™ 2000
- INO-4500 Group B (Experimental): Participants will receive 2 ID injections of 1 mg/dose INO-4500 followed by EP using the CELLECTRA™ 2000 device in two acceptable locations in two different limbs at each dosing visit.
  Interventions: Drug: INO-4500; Device: CELLECTRA™ 2000
- Placebo Group C (Placebo Comparator): Participants will receive 1 ID injection of 1 mg/dose placebo followed by EP using the CELLECTRA™ 2000 device.
  Interventions: Device: CELLECTRA™ 2000; Drug: Placebo
- Placebo Group D (Placebo Comparator): Participants will receive 2 ID injections of 1 mg/dose placebo followed by EP using the CELLECTRA™ 2000 device in two acceptable locations in two different limbs at each dosing visit..
  Interventions: Device: CELLECTRA™ 2000; Drug: Placebo

INTERVENTIONS:
Drug: INO-4500 — INO-4500 will be administered ID on Day 0 and Week 4.
  Arms: INO-4500 Group A; INO-4500 Group B
Device: CELLECTRA™ 2000 — EP using the CELLECTRA™ 2000 device will be administered following ID drug administration.
Drug: Placebo — Placebo will be administered ID on Day 0 and Week 4.
  Other Names: SSC-0001
  Arms: Placebo Group C; Placebo Group D

SUMMARY:
This is a randomized, blinded, placebo-controlled trial to evaluate the safety, tolerability and immunological profile of INO-4500 administered by intradermal (ID) injection followed by electroporation (EP) using CELLECTRA™ 2000 device in healthy volunteers in Ghana.

ELIGIBILITY:
Inclusion Criteria:

* Judged to be healthy by the Investigator on the basis of medical history, physical examination and vital signs performed at Screening;
* Negative tests for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody and Human Immunodeficiency Virus (HIV) antibody;
* Screening electrocardiogram (ECG) deemed by the Investigator as having no clinically significant findings (e.g. Wolff-Parkinson-White syndrome);
* Must meet one of the following criteria with respect to reproductive capacity: Surgically sterile or have a partner who is sterile (i.e., vasectomy in males or tubal ligation, absence of ovaries and/or uterus in females). In the case of vasectomy, participants should wait six (6) months post-vasectomy prior to enrolling. Women who are post-menopausal as defined by absence of menstruation for ≥ 12 months. Use of medically effective contraception when used consistently and correctly from Screening until three (3) months following last dose.

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant or father children within the projected duration of the trial starting with the screening visit until three (3) months following last dose;
* Positive serum pregnancy test during Screening or positive urine pregnancy test prior to any dosing;
* Is currently participating in or has participated in a study with an investigational product within 30 days preceding Day 0;
* Previous receipt of an investigational vaccine product for prevention of Lassa Fever;
* Audiometry testing that demonstrates a hearing level threshold greater than 30 dB for any frequency tested between 500 Hz - 8000 Hz;
* Fewer than two acceptable sites available for ID injection and EP considering the deltoid and anterolateral quadriceps muscles;
* Current or anticipated concomitant immunosuppressive therapy;
* Fever with or without cough or any other concurrent illness which the principal investigator feels is contraindicated to clinical trial participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Baseline up to Week 48
Number of Participants with Injection Site Reactions | Day 0 up to Week 48
Number of Participants with Adverse Events of Special Interest (AESIs) | Baseline up to Week 48
Change from Baseline in Lassa Virus (LASV) Antigen Specific Binding Antibodies | Day 0 up to Week 48
Change from Baseline in Lassa virus (LASV) Neutralization Assays | Day 0 up to Week 48
Change from Baseline in Interferon-Gamma Response Magnitude | Day 0 up to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Orizu, MD, Study Director — Inovio Pharmaceuticals
Locations (1):
- Noguchi Memorial Institute for Medical Research, University of Ghana, Legon, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to two (2) years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.

REFERENCES:
- [Derived] Koram KA, Walker KA, Orizu B, Marrero I, Boyer J, Yang S, Broderick KE, Kusi KA, Kyei-Baafour E, Ofori EA, Pobee A, Adu-Amankwah S, Amoakoh-Coleman M, Amoakoh HB, Abuaku B, Badji E, Ntiri M, Quaye L, Morrow MP, Sylvester AJ, Reuschel EL, Gillespie E, Liebowitz D, Humeau LM. Safety, tolerability, and immunogenicity of INO-4500, a synthetic DNA-based vaccine against Lassa virus, in a phase 1b clinical trial in healthy Ghanaian adults. Front Immunol. 2025 Oct 24;16:1658549. doi: 10.3389/fimmu.2025.1658549. eCollection 2025. PMID 41208990